CLINICAL TRIAL: NCT01743495
Title: CAPABLE for Frail Dually Eligible Older Adults
Acronym: CAPABLE500
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency); Baltimore City Health Department (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NA_00076471; 1C1CMS330970-01-00 (Other: Centers for Medicare and Medicaid Services)
Record Dates: First submitted 2012-10-15; First posted 2012-12-06 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Muscle Weakness
Keywords: Medical Costs; improved IADLs; and/or ADL's; decreased nursing home admissions
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Functional Services (Other): The program consists of up to 10 home-based functional services sessions over 4 months.
  Interventions: Behavioral: 10 home-based functional services sessions over 4 months.

INTERVENTIONS:
Behavioral: 10 home-based functional services sessions over 4 months. — The program consists of up to 10 home-based functional services sessions over 4 months.

SUMMARY:
The Johns Hopkins School of Nursing offers this research study which aims to learn more about whether services that help with medications, muscle strengthening, pain management and changes to houses can help improve older adults' ability to, walk, and take care of themselves while saving costs by reducing hospitalizations and nursing home admissions.

DETAILED DESCRIPTION:
* 65yrs or older
* Be able to stand (with or without assistance)
* Have some difficulty with getting dressed, or preparing food, bathing
* Receive a low monthly income
* Have no plans to move in the next year
* NOT be receiving home nursing or other therapy right now

ELIGIBILITY:
Inclusion Criteria:

* 65 or older
* Cognitively intact (≥ 10 on Brief Interview of Mental Status)
* Difficulty with ≥ 2 IADLS or ≥ 1 ADL
* ≤ 199% of Federal Poverty level

Exclusion Criteria:

* Terminally ill

  --Active cancer treatment
* Hospitalized > 3 times in last 3 years
* Receiving home nursing, Occupational Therapy or Physical Therapy
* Don't have phone or do plan to move in less than a year

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 281 (Actual)
Dates: Start 2012-09; Primary Completion 2018-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Cost Effective | one year after intervention
  Chart review to see change between cost of intervention to medicaid before and after CAPABALE
Cost Effective | two years after intervention
  Chart review to see change between cost of intervention to medicaid before and after CAPABALE
Cost Effective | one year after intervention
  Chart review to see change between cost of intervention to medicare before and after CAPABALE
Cost Effective | two years after intervention
  Chart review to see change between cost of intervention to medicare before and after CAPABALE

SECONDARY OUTCOMES:
Quality of Life as assessed by the Activities of Daily Living (ADL) Questionnaire | four months post intervention
  The ADL Questionnaire will be used to assess quality of life in participants. The score ranges from 0 to 32, with 0 being no help required with activities of daily life and 32 representing that the participant is incapable of completing activities of daily life regardless of difficulty without assistance.
Quality of Life as assessed by the ADL Questionnaire | eight months post intervention
  The ADL Questionnaire will be used to assess quality of life in participants. The score ranges from 0 to 32, with 0 being no help required with activities of daily life and 32 representing that the participant is incapable of completing activities of daily life regardless of difficulty without assistance.
Quality of Life as assessed by the ADL Questionnaire | twelve months post intervention
  The ADL Questionnaire will be used to assess quality of life in participants. The score ranges from 0 to 32, with 0 being no help required with activities of daily life and 32 representing that the participant is incapable of completing activities of daily life regardless of difficulty without assistance.
Quality of Life as assessed by the Instrumental Activities of Daily Living (IADL) Questionnaire | four months post intervention
  The IADL Questionnaire will be used to assess quality of life in participants. The score ranges from 0 to 32, with 0 being no help required with activities of daily life and 32 representing that the participant is incapable of completing instrumental activities of daily life regardless of difficulty without assistance.
Quality of Life as assessed by the IADL Questionnaire | eight months post intervention
  The IADL Questionnaire will be used to assess quality of life in participants. The score ranges from 0 to 32, with 0 being no help required with activities of daily life and 32 representing that the participant is incapable of completing instrumental activities of daily life regardless of difficulty without assistance.
Quality of Life as assessed by the IADL Questionnaire | twelve months post intervention
  The IADL Questionnaire will be used to assess quality of life in participants. The score ranges from 0 to 32, with 0 being no help required with activities of daily life and 32 representing that the participant is incapable of completing instrumental activities of daily life regardless of difficulty without assistance.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Szanton, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szanton SL, Alfonso YN, Leff B, Guralnik J, Wolff JL, Stockwell I, Gitlin LN, Bishai D. Medicaid Cost Savings of a Preventive Home Visit Program for Disabled Older Adults. J Am Geriatr Soc. 2018 Mar;66(3):614-620. doi: 10.1111/jgs.15143. Epub 2017 Nov 22. PMID 29165789
- [Derived] Waldersen BW, Wolff JL, Roberts L, Bridges AE, Gitlin LN, Szanton SL. Functional Goals and Predictors of Their Attainment in Low-Income Community-Dwelling Older Adults. Arch Phys Med Rehabil. 2017 May;98(5):896-903. doi: 10.1016/j.apmr.2016.11.017. Epub 2016 Dec 19. PMID 28007445